CLINICAL TRIAL: NCT06924073
Title: Scale-up of an Evidence-based Adolescent Transition Package to Support Transitional Care Among Youth Living With HIV
Acronym: ATTACH-Scale
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Kenyatta National Hospital (Other Government); University of Nairobi, Kenya (Unknown)
Responsible Party: Principal Investigator, Kristin Beima-Sofie, Senior Research Scientist, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00020373; 1R01MH136897 (NIH)
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Adolescent HIV Infection; Transition to Adult Care; Implementation Science; Implementation Strategies
Keywords: Adolescent HIV; Transition to Adult Care; Scale-up; Implementation science; implementation strategy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training of trainers (No Intervention): Sites assigned to the standard of care (SoC) control arm will receive cascading training of trainers (ToTs) and cascade training to sites for supporting scale-up of the ATP
- Youth Enhanced Implementation Strategy (ATP-YES) (Experimental): Sites assigned to the intervention arm will receive the ATP-YES implementation strategy, a multi-component youth led implementation strategy that incorporates data audits and feedback, cyclical small tests of change and learning collaboratives, to support scale-up of the ATP
  Interventions: Other: ATP-Youth Enhanced Strategy (ATP-YES)

INTERVENTIONS:
Other: ATP-Youth Enhanced Strategy (ATP-YES) — ATP-YES is a multi-component youth led implementation strategy that incorporates data audits and feedback, cyclical small tests of change and learning collaboratives
  Arms: Youth Enhanced Implementation Strategy (ATP-YES)

SUMMARY:
Ending the HIV epidemic for youth living with HIV will require implementation and optimization of evidence-based interventions that address barriers to treatment. The proposed implementation study will test a youth-led data-driven implementation strategy to scale-up an evidence-based Adolescent Transition Package (ATP) aimed at improving transition processes and post-transition clinical outcomes for youth living with HIV in Kenya. Clinics will be randomized to receive standard of care implementation through trainer of trainers or the youth-led data-driven implementation strategy alongside trainer of trainers. We will study whether the enhanced implementation strategy improves the number of youth who receive the ATP, the number of providers that initially chose to use the ATP, and the consistency with which the ATP is used over time. We will also evaluate the cost of the ATP and whether the ATP improves health outcomes among youth living with HIV, including viral suppression and retention in care. Healthcare workers at study sites will complete surveys, focus group discussions, interviews, and participate in continuous quality improvement processes. Youth will participate in surveys and focus groups, and have their routine medical records abstracted.

DETAILED DESCRIPTION:
The proposed project extends the team's previously conducted cluster randomized controlled trial, the Adolescent Transition to Adult Care (ATTACH) study (NIH R01HD089850-01; PI John-Stewart). This new R01 tests an implementation strategy to improve scale up of an Adolescent Transition Package (ATP), developed during the previous clinical trial, within health facilities in Kenya and evaluate the cost-effectiveness and budget impact of the implementation strategy. Primary outcomes include measuring intervention uptake and delivery outcomes using the Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) framework, factors influencing implementation, clinical outcomes, and cost.

The ATP is a healthcare worker (HCW) delivered toolkit that supports the transition from pediatric to independent care for youth living with HIV (YLH). The ATP was developed by the ATTACH study, working in partnership with the Kenya Ministry of Health and other key collaborators leading treatment and care provision in Kenya. The ATP is designed to support transition to adult care for YLH and provide YLH with the knowledge and skills needed to independently manage HIV. The ATP combined two evidence-based interventions from other contexts (Namibia and the United States) and adapted them to better meet Kenyan patient, provider and health system needs. The ATP was tested in a randomized controlled trial of 20 clinics in 4 counties in Kenya (ATTACH study), and shown to significantly improve readiness to transition among YLH in intervention sites compared to those in the control. HCWs and YLH appreciated the content and design of the ATP as they found it feasible and acceptable for routine clinic use.

During this scale up focused R01, the ATP will be administered at the clinic level by existing HCWs during routine YLH clinic visits, as in the original trial. In all participating clinics, all eligible adolescents aged 10-24 years will have medical record data abstracted, and older YLH (ages 15-24) will be offered the opportunity to participate in surveys and qualitative data collection. HCWs from participating clinics will provide feedback on implementation throughout the study and work to optimize delivery of the ATP within their clinic settings.

The ATTACH-Scale study includes implementation of the ATP in 32 clinics. The 32 study sites for this R01 will be selected from a large list of eligible facilities, and specific clinics will be selected by prioritizing high HIV volume clinics (>50 YLH per clinic), existing collaborations (ex: ATTACH study sites), and MoH priorities. Selection of intervention and control sites will be done using stratified randomization, balancing for county and model of HIV care in the clinic, by a biostatistician based at the University of Washington. The units of analysis vary by study aim, and are either at the level of the HCW, YLH, or clinic, depending on the specific aim and outcome being assessed.

Specific details for each study aim are described below.

Aim 1 (SCALE-UP): Using an effectiveness-implementation hybrid III design, the study will test the impact of ATP scale-up using the Kenya MoH standard of care (SoC) implementation strategy (Trainer of Trainers [ToT]) versus an enhanced scale-up implementation strategy that includes the SoC plus youth-led data- driven intervention adaptations (ATP-YES). ATP-YES is a multi-component youth led package that incorporates weekly data assessments, data review and adaptation meetings, and cross collaborative learning across intervention sites. In total, 32 HIV clinics (4 counties, 8 per county) will be randomized 1:1 to 36 months of ATP-YES or SoC alone. The Reach, Effectiveness, Adoption, Implementation and Maintenance [RE-AIM] framework will be used to evaluate and compare ATP implementation and guide real-time ATP adaptations. Specifically, ATP reach (YLH exposed to ATP), effectiveness (intervention effect on transition readiness, viral suppression and retention), adoption (proportion of HCWs implementing the ATP), implementation (fidelity to ATP processes), and maintenance (continued use post-trial) will be measured at each study site and compared between intervention and control arms. The Consolidated Framework for Implementation Research (CFIR) will be used to understand the role of context on how and why the ATP-YES strategy is or is not successful. The Framework for Reporting Adaptations and Modifications to Evidence-based Implementation Strategies (FRAME-IS) will be used to systematically study adaptations to the ATP and ATP-YES implementation strategy.

Aim 2 (COSTING): Simultaneously with Aim 1, program costs will be captured and the budget impact of ATP-YES will be compared between intervention and control sites. Micro costing, involving HCW interviews and time and motion observations, will be used to estimate the incremental costs of implementing the ATP-YES strategy and develop a model to project the health impact (HIV deaths and morbidity averted) and financial costs of ATP-YES compared to SoC.

Impact: The study will determine whether the ATP-YES can be used to effectively and affordably support implementation of the ATP in Kenya. The study team hypothesizes that this implementation strategy will improve uptake, integration, and delivery of the ATP within existing YLH clinics.

Alongside study aims, this project will engage communities, build capacity for IS research among youth, program implementers and policy-makers, and participate in collaborative science. The project includes collaboration with MOH in Kenya to ensure transition tools and implementation processes align with and integrate MOH priorities and strategies. The study also includes creation of a youth advisory board and engagement of policy-makers, HCWs, program implementers and other key stakeholders throughout the entirety of the study. Finally, the study supports youth to gain research skills and build capacity for conducting research through their leadership roles in ATP-YES, involvement in youth mentorship programs, and the youth advisory board.

ELIGIBILITY:
Inclusion Criteria:

Healthcare providers

* ≥18 years of age
* Employed at one of the 32 facilities in the RCT
* Provides HIV services to adolescents affiliated within their clinic Adolescents and youth living with HIV
* Between 15-24 years of age (focus group discussions, surveys) or between 10-24 years of age (offered the intervention)
* Receives HIV clinical care at one of the clinics included in the study
* Attended clinic ≥1 time following intervention implementation

Exclusion Criteria:

Any individual who meets the following criteria will be excluded from participation in this study:

- Conditions that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1920 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2029-01-30 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
Reach | From enrollment through 6 months post study end (42 months)
  Proportion of youth living with HIV ages 15-24 years exposed to the ATP intervention
Effectiveness: Successful Transfer | From enrollment through 6 months post study end (42 months)
  Proportion of youth living with HIV who attend first adult clinic visit
Effectiveness: Retention | From enrollment through 6 months post study end (42 months)
  Number of scheduled clinic visits youth living with HIV attend in the year after transition to adult care
Adoption | From enrollment through 6 months post study end (42 months)
  Proportion of health providers in youth HIV clinics who deliver the ATP

SECONDARY OUTCOMES:
Effectiveness: Transition Readiness | From enrollment through 6 months post study end (42 months)
  Change in transition readiness scores
Effectiveness: Viral Suppression | From enrollment through 6 months post study end (42 months)
  Proportion of youth living with HIV who are virally suppressed 12 months after transition to adult clinics
Implementation: Fidelity to ATP | From enrollment through 6 months post study end (42 months)
  Proportion of facilities that deliver the ATP as designed
Implementation: Fidelity to ATP-YES | From enrollment through 6 months post study end (42 months)
  Proportion of facilities that deliver the ATP-YES as designed in intervention clinics
Maintenance | From study end (36 months) through 6 months post study end (42 months)
  Proportion of clinics that continue use the ATP as designed 6 months post study

OTHER OUTCOMES:
Reach | From enrollment through 6 months post study end (42 months)
  Proportion of YLH who do not know their HIV status who are exposed to the disclosure intervention
Effectiveness: Disclosure | From enrollment through 6 months post study end (42 months)
  Proportion of YLH who know their HIV status

CONTACTS AND LOCATIONS:
Overall Officials: Kristin M Beima-Sofie, PhD, MPH, Principal Investigator — University of Washington; Irene Njuguna, MBChB, MPH, PhD, Principal Investigator — Kenyatta National Hospital; Grace John-Stewart, MD, PhD, MPH, Principal Investigator — University of Washington; Dalton Wamalwa, MBChB, MMed, MPH, Principal Investigator — University of Nairobi
Locations (25):
- Kenya (25):
  - Awendo Sub County Hospital, Awendo
  - Uriri Sub County Hospital, Awendo
  - Gatundu Level 5 Hospital, Gatundu
  - Kiambu County Referral Hospital, Kiambu
  - Wangige Sub-County Hospital, Kiambu
  - Kikuyu (PCEA) Hospital, Kikuyu
  - Nazareth Hospital, Limuru
  - Arombe Dispensary, Migori
  - Dede Health Centre, Migori
  - Migori County Referral Hospital, Migori
  - St Joseph Mission Hospital (Ombo), Migori
  - Baraka Dispensary (Nairobi), Nairobi
  - Embakasi Health Centre, Nairobi
  - Kenyatta National Hospital/University of Nairobi, Nairobi
  - Mama Lucy Kibaki Hospital, Nairobi
  - Mbagathi District Hospital, Nairobi
  - Mukuru Health Centre, Nairobi
  - Pumwani Maternity Hospital, Nairobi
  - Tabitha Medical Clinic, Nairobi
  - Umoja Health Center, Nairobi
  - Rongo Sub County Hospital, Rongo
  - Verna Health Centre, Rongo
  - Ruiru Sub-County Hospital, Ruiru
  - Kiandutu Health Centre, Thika
  - Thika Level 5 Hospital, Thika

IPD SHARING:
Plan to Share IPD: Yes
The research community will have access to data when the award ends. De-identified individual and aggregate survey data (including raw and recoded data) will be deposited to NDA starting 12 months after the award begins and will be deposited every six months thereafter following the usual NDA data submission dates. As required by NDA, studies will also be created that contain the data used for every publication.
  Documentation to be made publicly available to the research community will include PDF, Word, and Excel documents containing survey instruments, interview guides, data collection protocols, codebooks for surveys and qualitative analysis, and code used in survey data analyses.
  Abstracted medical records will be used as secondary data and will not be shared. Transcripts from focus group discussions and interviews with providers, and voice recordings of focus groups or interviews from youth and providers will not be shared to protect participant privacy.